CLINICAL TRIAL: NCT03777215
Title: Angiotensin-(1-7) and Energy Expenditure in Human Obesity
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Amy Arnold (Other)
Responsible Party: Sponsor-Investigator, Amy Arnold, Associate Professor, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 9895
Record Dates: First submitted 2018-12-12; First posted 2018-12-17 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — angiotensin I (1-7); Acetates; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Angiotensin-(1-7) (Experimental): Subjects will receive intravenous infusion of three ascending doses of angiotensin-(1-7). The doses are: 2, 4, and 8 ng/kg/min. Each dose will be maintained for 10 minutes, with the highest dose maintained for an additional 90 minutes. The total infusion period is 120 minutes.
  Interventions: Drug: Angiotensin-(1-7)
- Placebo (Placebo Comparator): Subjects will receive intravenous infusion of saline that is matched in volume to the angiotensin-(1-7). The total infusion period is 120 minutes.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Angiotensin-(1-7) — This is a biologically active beneficial hormone of the renin-angiotensin system.
  Other Names: Angiotensin I/II (1-7) Acetate
  Arms: Angiotensin-(1-7)
Drug: Saline — Saline will be used as the placebo comparator.
  Other Names: 0.9% sodium chloride; normal saline
  Arms: Placebo

SUMMARY:
The objective of this study is to better define the role of the hormone angiotensin-(1-7) in energy balance. We will test the overall hypothesis that angiotensin-(1-7) increases resting energy expenditure and promotes markers of heat production (thermogenesis) in white adipose tissue in human obesity.

DETAILED DESCRIPTION:
Angiotensin-(1-7) is a beneficial hormone of the renin-angiotensin system known to produce positive cardiovascular and metabolic effects in animal models. In this study, the investigators will determine if angiotensin-(1-7) can increase resting energy expenditure and promote white adipose tissue heat production (thermogenesis) in obese human subjects. The investigators will perform a randomized, double-blind, two-arm parallel group study to determine effects of acute intravenous angiotensin-(1-7) versus saline infusion on resting energy expenditure measured by indirect calorimetry in obese human participants. In addition, blood pressure and heart rate will be measured and blood samples obtained to measure for changes in circulating renin-angiotensin system and metabolic hormones. Abdominal subcutaneous white adipose biopsies will also be obtained from obese human participants during acute angiotensin-(1-7) versus saline infusions to examine for changes in gene expression for markers of thermogenesis. The findings from these studies will advance understanding of hormonal mechanisms involved in the etiology of obesity, and provide new insight into the potential for targeting angiotensin-(1-7) to improve energy balance in human obesity.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of all races
* Capable of giving informed consent
* Age 18-60 years
* Body mass index (BMI) between 30-40 kg/m2
* Satisfactory history and physical exam

Exclusion Criteria:

* Age ≤ 17 or ≥ 61 years
* Pregnant, nursing, or postmenopausal women
* Decisional impairment
* Prisoners
* Alcohol or drug abuse
* Current smokers
* Highly trained athletes
* Claustrophobia
* Subjects with >5% weight change in the past 3 months
* Evidence of type I or type II diabetes (fasting glucose > 126 mg/dL or use of anti-diabetic medications)
* History of serious cardiovascular disease other than hypertension (e.g. myocardial infarction within 6 months, symptomatic coronary artery disease, presence of angina pectoris, significant arrhythmia, congestive heart failure, deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis, hypertrophic cardiomyopathy) or cerebrovascular disease (e.g. cerebral hemorrhage, stroke, transient Ischemic attack).
* History or presence of immunological or hematological disorders
* Impaired hepatic function (aspartate aminotransferase or alanine aminotransferase levels >2 times upper limit of normal range)
* Impaired renal function (serum creatinine >2.0 mg/dl)
* Anemia
* Treatment with anticoagulants (e.g. warfarin)
* Treatment with chronic systemic glucocorticoid therapy (>7 consecutive days in 1 month)
* Treatment with medications influencing energy expenditure (e.g. psychostimulants)
* Treatment with any investigational drug in the 1-month preceding the study
* Inability to give, or withdraw, informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Resting energy expenditure | 120 minutes
  Change in resting energy expenditure measured by indirect calorimetry at baseline and at end of angiotensin-(1-7) versus saline infusion.
Uncoupling protein 1 | 120 minutes
  White adipose tissue biopsies will be taken at end of angiotensin-(1-7) versus saline infusion to assess gene expression of the heat producing (thermogenic) marker uncoupling protein 1.

SECONDARY OUTCOMES:
Blood pressure | 120 minutes
  Change in arm and finger cuff blood pressure following angiotensin-(1-7) versus saline infusion
Heart rate | 120 minutes
  Change in heart rate following angiotensin-(1-7) versus saline infusion

OTHER OUTCOMES:
Skin temperature | 120 minutes
  Change in skin temperature following angiotensin-(1-7) versus saline infusion
Skin blood flow | 120 minutes
  Change in skin blood flow following angiotensin-(1-7) versus saline infusion
Abdominal heat production | 120 minutes
  Change in abdominal heat production as measured by thermal imaging following angiotensin-(1-7) versus saline infusion
Catecholamines | 120 minutes
  Change in plasma catecholamines following angiotensin-(1-7) versus saline infusion
Insulin | 120 minutes
  Change in plasma insulin levels following angiotensin-(1-7) versus saline infusion
Glucose | 120 minutes
  Change in plasma glucose levels following angiotensin-(1-7) versus saline infusion
Fatty acids | 120 minutes
  Change in plasma free fatty acid levels following angiotensin-(1-7) versus saline infusion
Angiotensin II | 120 minutes
  Change in plasma angiotensin II levels following angiotensin-(1-7) versus saline infusion
Angiotensin-(1-7) | 120 minutes
  Change in plasma angiotensin-(1-7) levels following angiotensin-(1-7) versus saline infusion
Renin | 120 minutes
  Change in plasma renin activity following angiotensin-(1-7) versus saline infusion
Aldosterone | 120 minutes
  Change in plasma aldosterone levels following angiotensin-(1-7) versus saline infusion

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Arnold, PhD, Principal Investigator — Pennsylvania State University College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.